CLINICAL TRIAL: NCT04729985
Title: Daibetes Discharge Transitional CGM Study
Brief Title: Diabetes Discharge Transitional CGM Study (DDT-CGM)
Acronym: DDT-CGM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Christopher Jones, Principal Investigator, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1051438
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: hospital discharge; Continuous Glucose Monitoring; Type 2 diabetes; rehospitalization
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Trial
Who Masked: Outcomes Assessor
Masking Description: Data evaluation group will be blinded as to which arm the data comes from
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Care (No Intervention): A blinded CGM will be placed to review glucoses after discharge in the Standard Care arm.
- Diabetic education and CGM monitoring (Active Comparator): Treatment arm will get diabetic education, active CGM use with patient feedback for 14 days, active access to the PI for concerns relating to hospitalization. They will also receive a brief, 15 minute phone call from the PI on day 3-4, 6-7, 9-10 and day 14-15.
  Interventions: Device: CGM device with diabetic education, CGM education and a follow up protocol.

INTERVENTIONS:
Device: CGM device with diabetic education, CGM education and a follow up protocol. — Blind CGM placed and recorded for 14 days after discharge and data downloaded
  Other Names: Blind CGM
  Arms: Diabetic education and CGM monitoring

SUMMARY:
Intervention group will receive brief diabetic education, CGM education and use and have a CGM placed before discharge. They will also sign up for "Cloud" access of their CGM data. A medical assistant will review their CGM data daily to make sure they are using the CGM adequately. The principal investigator will review the CGM data and call the patient for a brief phone evaluation of their glucoses and their transition from the hospital to outpatient care. The will be called 4 times between discharge and day 15 by the principal investigator.

Standard treatment group will receive a blinded CGM to be reviewed 30 days after discharge.

Reduction in hospitalizations and ER visits within the first 30 days is the primary outcome. Time in range, hypoglycemia, hyperglycemia and patient satisfaction will also be evaluated 30 days after discharge.

DETAILED DESCRIPTION:
Patients admitted to a community hospital with diabetes will be evaluated for being high risk for rehospitalization. High risk patients will be identified and those that are found to be high risk will be evaluated for entrance to the study and consented.

Those that consent will be randomized to two arms, an intervention arm and a standard care arm with CGM monitoring.

Intervention will include a brief 15 minute diabetic education session and a 15 minute brief education on how to use the Freestyle Libre CGM. A sensor will be placed and initiated before discharge. They will also sign up for a Freestyle Libre View account and grant access to the intervention team. The will receive a handout of reasons to call the principal investigator during the first 15 days and will be told to access the PI through the hospital operator. The PI will call the patient on day 3-4, day 5-6, day 9-10 and day 14-15 after reviewing their CGM data. The PI will review their glucoses and also any concerns from their hospitalization. The team can then help bridge any treatment or care gaps with the patients PCP or care team. The CGM data will be recorded for the first 14 days and data will be sent to the PCP.

The standard treatment arm will get 15 minutes of education on how to use the Libre Pro blinded CGM sensor and the sensor will be placed before discharge. The sensor will be sent back the the team and downloaded. After 30 days the data will be sent to the patients PCP.

Outcomes will be measured for 30 days from discharge.

Patient satisfaction will be measured by a phone interview in both groups once after 31-40 days from discharge

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes plus one additional criteria during hospitalization:

A1C greater than or equal to 9, New diagnosis of diabetes Type 2 and A1C greater than or equal to 8, On insulin, On sulfonylurea, Deemed to by high risk by hospitalist staff for post-hospitalization complications, Acute Heart Failure, Acute Coronary Syndrome (ACS), Stroke, or a TIA.

-

Exclusion Criteria:

Type 1 Diabetes, or Not high risk (as above), or Already using a CGM, or Unable to understand or use a CGM, or Unable or unwilling to use a CGM, or Participating in another clinical trial within 30 days.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Emergency room visit and rehospitalization | Within 30 days after discharge from the hospital
  Total Emergency room visits and total rehospitalizations

SECONDARY OUTCOMES:
Emergency room visits | Within 30 days after discharge from the hospital
  Total Emergency room visits
Rehospitalizations | Within 30 days after discharge from the hospital
  Total Rehospitalizations
Time in range | From discharge to day 14
  percent of time glucose is in range from 70-180 mg/dl as measured by CGM
time in hypoglycemia | from discharge through day 14
  amount of time below 70 mg/dl as measured by CGM
Severe hypoglycemia | from discharge to day 30
  hypoglycemia requiring the assistance from another person
time in hyperglycemia | From discharge through day 14
  glucose from 181-250 mg/dl as measured by CGM
time in severe hyperglycemia | from discharge through day 14
  glucose greater than 251 mg/dl as measured by CGM
Patient satisfaction | survey will be done between 31 and 40 days after hospital discharge
  Patient telephone questionnaire about patient satisfaction during the transition phase

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Jones, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Logan Regional Hospital, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No